CLINICAL TRIAL: NCT07112547
Title: Occurrence of Severe Cardiac Rhythm and Conduction Disturbances in Emergency Department Patients With Non-ST Elevation Acute Coronary Syndrome
Acronym: SurvSCA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9460
Record Dates: First submitted 2025-05-27; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Coronary Syndrome Without ST Elevation on Electrocardiogram; Acute Coronary Syndromes (ACS); Myocardial Infarction, Unstable Angina Pectoris, Sudden Cardiac Death, Stroke, Peripheral Artery Disease
Keywords: Non-ST Segment Elevation Acute Coronary Syndrome; Cardiac Arrhythmias; Heart Conduction System Disease; Hospital Emergency Service; Electrocardiographic monitoring; Cardiovascular diseases
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable; Death, Sudden, Cardiac; Stroke; Peripheral Arterial Disease; Arrhythmias, Cardiac; Emergencies; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-ST segment elevation ACS: 500 adult patients admitted to the emergency department and diagnosed with non-ST segment elevation ACS

SUMMARY:
Cardiovascular diseases are the leading cause of death worldwide. Among them, coronary artery disease-especially in its acute form, known as acute coronary syndrome (ACS)-is the most frequent cause of cardiovascular death. There are two main types of ACS: ST-segment elevation myocardial infarction (STEMI) and non-ST-segment elevation ACS (NSTE-ACS). While the occurrence of serious heart rhythm and conduction disturbances is well established in STEMI, these complications are believed to be much less frequent in NSTE-ACS. However, their actual frequency in this population remains unclear due to limited studies, especially in emergency settings.

The main purpose of this study is to estimate the frequency of serious rhythm and conduction disorders in patients presenting with NSTE-ACS in emergency departments. The hypothesis is that these events are rare in this population and may not justify routine continuous cardiac monitoring for all such patients, as currently recommended.

Secondary objectives include identifying risk factors for these complications, estimating their frequency during hospitalization, assessing the frequency of minor rhythm and conduction disorders, evaluating care times and patient flow in emergency departments, and assessing patient outcomes up to 30 days-including hospitalizations, length of stay, discharge disposition, all-cause mortality, and the occurrence of five major adverse cardiovascular events (5-point MACE).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old) patient admitted to the emergency department
* Able to understand the information provided
* Diagnosis of non-ST segment elevation ACS established according to the lastest guidelines from the European Society of Cardiology and the 4th Universal Definition of myocardial infarction
* No objection to participation in the study after receiving appropriate information

Exclusion Criteria:

* Patients subject to legal protection
* Patient with cognitive impairment
* Myocardial injury and/or symptoms attributable to Takotsubo syndrome, myocarditis, pericarditis, or acute heart failure
* Clinical evidence suggestive of type 2 myocardial infarction, including acute anemia with hemoglobin < 10 g/dL, sepsis, acute hypoxemic respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the emergency department and diagnosed with non-ST segment elevation ACS
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Serious Rhythm or Conduction Disturbances in the Emergency Department | During emergency department stay, assessed up to 24 hours
  Occurrence of at least one serious rhythm or conduction disturbance during emergency department management, including: sustained ventricular tachycardia (VT), ventricular fibrillation (VF), torsades de pointes, high-degree conduction disorders (Mobitz type II AV block, third-degree AV block, trifascicular block), pulseless electrical activity (PEA), and asystole.

SECONDARY OUTCOMES:
Incidence of Non-Life-Threatening Arrhythmias or Conduction Disorders in the Emergency Department | During emergency department stay, assessed up to 24 hours
  Occurrence of arrhythmias not immediately life-threatening: atrial fibrillation or flutter, Mobitz type I AV block, first-degree AV block, sinus node dysfunction, or non-sustained VT
Number of patients presenting complications prior to a confirmed diagnosis of NSTE-ACS | Prior to establishing a confirmed diagnosis of NSTE-ACS in the ED, assessed up to 12 hours
  Occurrence of complications such as syncope, presyncope, cardiogenic shock, respiratory distress, or rhythm/conduction disturbances before final diagnosis of NSTE-ACS.
Duration of Stay in the Emergency Department | From ED admission to hospital admission, discharge, or UHCD discharge; up to 72 hours
  Time spent in the emergency department and in the short-stay unit (UHCD) before transfer or discharge.
Number of patients by disposition at emergency department discharge (home vs. hospital admission and type of admitting service | At the time of emergency department discharge or transfer, assessed up to 72 hours from ED admission
  Disposition of patients: home discharge or hospital admission. For admitted patients, type of service recorded (ICU, coronary care unit, cardiology, internal medicine, short-stay unit, or other).
Duration of Hospitalization | From hospital admission to hospital discharge, assessed up to 14 days.
  Overall length of stay for hospitalized patients
Number of patients with all-cause mortality or 5-point major adverse cardiovascular events (5P-MACE) at 30 days | Day 30 post-ED management
  This composite outcome includes the number of participants who experience either all-cause death or at least one of the following 5-point major adverse cardiovascular events (5P-MACE) within 30 days:
  1. Cardiovascular death
  2. Myocardial infarction
  3. Stroke or transient ischemic attack (TIA)
  4. Hospitalization for heart failure
  5. Coronary or peripheral revascularization Outcome events will be assessed through medical records and/or follow-up phone call if needed.
Clinical features : weight | From admission to discharge from hospital, assessed up to 7 days
  Weight (kg)
Clinical features : height | From admission to discharge from hospital, assessed up to 7 days
  Height (cm)
Clinical features : heart rate | From admission to discharge from hospital, assessed up to 7 days
  Heart rate (bpm)
Clinical data : blood and arterial pressure | From admission to discharge from hospital, assessed up to 7 days
  systolic/diastolic blood pressure (mmHg) and mean arterial pressure (mmHg)
Clinical data : oxygen saturation | From admission to discharge from hospital, assessed up to 7 days
  peripheral capillary oxygen saturation (%)
Clinical data : temperature | From admission to discharge from hospital, assessed up to 7 days
  Temperature (°C)
clinical data : capillary blood glucose | From admission to discharge from hospital, assessed up to 7 days
  Capillary blood glucose g/L
Cardiovascular history and risk factors | From admission to discharge from hospital, assessed up to 7 days
  Cardiovascular history and risk factors : questionnaire on medical history and prior related treatments (anticoagulant, antiplatelet agent, analgesic, oxygen therapy, statin, beta blocker, ACE inhibitor, angiotensin II receptor blocker).
Biological workup : troponin | From admission to discharge from hospital, assessed up to 7 days
  Troponin (1st, 2nd ; 3rd measurement) (ng/mL)
Biological work-up : NT-proBNP | From admission to discharge from hospital, assessed up to 7 days
  NT-proBNP (ng/mL)
Biological workup : hemoglobin | From admission to discharge from hospital, assessed up to 7 days
  hemoglobin (g/dL)
Biological workup : BNP | From admission to discharge from hospital, assessed up to 7 days
  BNP (ng/mL)
Biological workup : platelets count | From admission to discharge from hospital, assessed up to 7 days
  platelets (10^9/L or Giga/L)
Biological workup : mean corpuscular volume | From admission to discharge from hospital, assessed up to 7 days
  mean corpuscular volume (fL or µm3)
Biological workup : potassium | From admission to discharge from hospital, assessed up to 7 days
  potassium (mmol/L)
Biological workup : creatinine | From admission to discharge from hospital, assessed up to 7 days
  creatinine (µmol/L)
Biological workup : creatinine clearance | From admission to discharge from hospital, assessed up to 7 days
  creatinine clearance (mL/min/1,73m2)
Electrocardiogram (ECG) | From admission to discharge from hospital, assessed up to 7 days
  Electrocardiogram (ECG) : presence or absence of ST elevation, T wave inversion, pathological

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina GARNIER-KEPKA, Dr, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (10):
- France (10):
  - Centre Hospitalier de Haguenau, Haguenau, Bas-Rhin
  - Centre Hospitalier de Sélestat, Séléstat, Bas-Rhin
  - Hôpitaux Universitaires de Strasbourg (NHC), Strasbourg, Bas-Rhin
  - Hôpital Louis Pasteur, Colmar, Haut-rhin
  - Hôpital Emilie Muller, Mulhouse, Haut-rhin
  - Hôpital Maison Blanche, Reims, Marne
  - CHRU de Nancy, Nancy, Meurthe-et-Moselle
  - Centre Hospitalier de Pont-à-Mousson, Pont-à-Mousson, Meurthe-et-Moselle
  - Centre Hospitalier de Toul Saint-Charles, Toul, Meurthe-et-Moselle
  - CHU de Poitiers, la Milétrie, Poitiers, Vienne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bouisset F, Ruidavets JB, Dallongeville J, Moitry M, Montaye M, Biasch K, Ferrieres J. Comparison of Short- and Long-Term Prognosis between ST-Elevation and Non-ST-Elevation Myocardial Infarction. J Clin Med. 2021 Jan 7;10(2):180. doi: 10.3390/jcm10020180. PMID 33430516
- [Background] Pines JM, Pollack CV Jr, Diercks DB, Chang AM, Shofer FS, Hollander JE. The association between emergency department crowding and adverse cardiovascular outcomes in patients with chest pain. Acad Emerg Med. 2009 Jul;16(7):617-25. doi: 10.1111/j.1553-2712.2009.00456.x. Epub 2009 Jun 22. PMID 19549010
- [Background] Timmis A, Vardas P, Townsend N, Torbica A, Katus H, De Smedt D, Gale CP, Maggioni AP, Petersen SE, Huculeci R, Kazakiewicz D, de Benito Rubio V, Ignatiuk B, Raisi-Estabragh Z, Pawlak A, Karagiannidis E, Treskes R, Gaita D, Beltrame JF, McConnachie A, Bardinet I, Graham I, Flather M, Elliott P, Mossialos EA, Weidinger F, Achenbach S; Atlas Writing Group, European Society of Cardiology. European Society of Cardiology: cardiovascular disease statistics 2021. Eur Heart J. 2022 Feb 22;43(8):716-799. doi: 10.1093/eurheartj/ehab892. PMID 35016208
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Glob Heart. 2018 Dec;13(4):305-338. doi: 10.1016/j.gheart.2018.08.004. Epub 2018 Aug 25. No abstract available. PMID 30154043
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Rev Esp Cardiol (Engl Ed). 2021 Jun;74(6):544. doi: 10.1016/j.rec.2021.05.002. No abstract available. English, Spanish. PMID 34020768